CLINICAL TRIAL: NCT06342518
Title: Clinical and Sonographic Evaluation of the Effectiveness of Extracorporeal Shock Wave Therapy (ESWT) in Patients With Lateral Epicondylitis
Brief Title: ESWT in Lateral Epicondylitis: Clinical,Ultrasonographic Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, MD, Specialist of PMR,Principal Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MU ESWT
Record Dates: First submitted 2024-03-24; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Lateral Epicondylitis; Tennis Elbow
Keywords: Extracorporeal Shock Wave Therapy (ESWT); sonographic assessment; Lateral epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Extracorporeal Shockwave Therapy; Exercise; Ice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT GROUP (Experimental): The ESWT group received radial ESWT on the painful lateral epicondyle once per week for a total of 3 sessions.
  A wrist resting splint, wrist extensor strengthening and stretching exercises, and ice treatment were administered to both groups.
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT); Behavioral: Resting Splint , Exercises and ice
- Sham-ESWT group (Sham Comparator): The Sham-ESWT group received Sham radial ESWT on the painful lateral epicondyle once per week for a total of 3 sessions.
  A wrist resting splint, wrist extensor strengthening and stretching exercises, and ice treatment were administered to both groups.
  Interventions: Device: Sham ESWT; Behavioral: Resting Splint , Exercises and ice

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy (ESWT) — The ESWT group received radial ESWT each session with a total of 2000 pulses at a frequency of 10 Hz. A gel was used at the interface, and the air pressure was set at 1.8 bar per session.
  Arms: ESWT GROUP
Device: Sham ESWT — The Sham-ESWT group received Sham radial ESWT each session, but without actual contact of the applicator. To enhance the illusion of treatment, gel was applied, and the device emitted sound at every shock
  Arms: Sham-ESWT group
Behavioral: Resting Splint , Exercises and ice — Ensuring proper usage of the wrist resting splint by the patient was confirmed during follow-up visits. The physician instructed the patients on stretching and strengthening exercises for wrist extensors, which they were asked to perform three times a day. Application of ice for 20 minutes every 3-4 hours during painful periods was recommended. During follow-up visits patients confirmed that they adherence to exercises and recommendations.

SUMMARY:
This study aimed to check and compare how well shock wave therapy works for tennis elbow, both in terms of symptoms and what we can see on ultrasound.

DETAILED DESCRIPTION:
42 patients with tennis elbow were split into two groups by chance: one group received shock wave therapy (ESWT), while the other received a fake treatment (Sham-ESWT) for comparison. Both groups underwent wrist exercises, splint usage, and ice application. Grip strength, pain levels, and how well they could move their wrist (functionality) were measured before, after, and one month post-treatment using tests. Additionally, the thickness of a common extensor tendon (CET) was evaluated using ultrasound. The patient, the doctor checking the patient, and the doctor doing the ultrasound didn't know which group the patient was in.

ELIGIBILITY:
Inclusion Criteria:

* experiencing pain and tenderness in the lateral epicondyle while extending their wrist and fingers against resistance for at least 3 months

Exclusion Criteria:

* Patients who are pregnant or have a coagulation disorder, cervical radiculopathy, peripheral neuropathy, peripheral vasculopathy in the upper extremity, complex regional pain syndrome, local infections, systemic inflammatory disease, fibromyalgia syndrome, arthritis (including rheumatoid arthritis, spondylarthritis, and crystal-induced arthropathies), malignancy, or those who have been treated with corticosteroids, PRP, or autologous blood injection, as well as those who have received physical therapy agents, undergone upper-extremity surgical interventions, or have a history of direct trauma to the elbow or a history of fracture,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Hand Grip Strength | Baseline, post-treatment(4th week), and one-month post-treatment (8th week)
  measured using the Jamar hand dynamometer
Pain severity | Baseline, post-treatment(4th week), and one-month post-treatment (8th week)
  Visual Analog Scale (VAS) which was scored from 0 (no pain) to 10 (extremely severe).
Functionality | Baseline, post-treatment(4th week), and one-month post-treatment (8th week)
  the Patient-Rated Tennis Elbow Evaluation (PRTEE)
  The PRTEE allows patients to rate their levels of tennis elbow pain and disability from 0 to 10, and consists of 2 subscales:
  1. PAIN subscale (0 = no pain, 10 = worst imaginable) Pain - 5 items
  2. FUNCTION subscale (0 = no difficulty, 10 = unable to do) Specific activities - 6 items Usual activities - 4 items In addition to the individual subscale scores, a total score can be computed on a scale of 100 (0 = no disability).
  Pain Score = Sum of the 5 pain items(out of 50) Best Score = 0, Worst Score =50 Function Score = Sum of the 10 function items, Divided by 2 (out of 50) Best Score = 0, Worst Score = 50
  Computing the Total Score Total Score = Sum of pain + function scores Best Score = 0, Worst Score = 50 Best Score = 0, Worst Score = 100
Quality of life score | Baseline, post-treatment(4th week), and one-month post-treatment (8th week)
  Short Form-12 (SF-12), Patients are provided with the SF-12 questionnaire, which consists of 12 questions covering physical and mental health domains.
  The scoring yields two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
  PCS mean score: 56,5 MSC mean score: 60.7 Scores above mean indicate a better-than-average health-related quality of life, while scores below mean suggest below-average health.
deep muscular tissue sensitivity | Baseline, post-treatment(4th week), and one-month post-treatment (8th week)
  pain pressure threshold (PPT) Pain pressure threshold (PPT) is used to measure deep muscular tissue sensitivity. The test determines the amount of pressure over a given area in which a steadily increasing nonpainful pressure stimulus turns into a painful pressure sensation. A varying pressure is applied from 0.5 to 1 kg/sec in a perpendicular direction relative to the muscle.
thickness of the common extensor tendon (CET) | Baseline, post-treatment(4th week), and one-month post-treatment (8th week)
  During ultrasonography for LE, the elbow is positioned in 90 degrees of flexion and the wrist in pronation. The ultrasound probe is placed longitudinally on the radial surface of the elbow. And common extensor tendon thickness was measured sonographically.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Physical Medicine and Rehabilitation Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No